CLINICAL TRIAL: NCT07293286
Title: Effect of Different Oxygen Concentrations During the Recovery Period Before Extubation After General Anesthesia on Hypoxemia After Extubation in Post-anesthesia Care Unit
Brief Title: Effect of Different Oxygen Concentrations Before Extubation After General Anesthesia on Hypoxemia After Extubation in Post-anesthesia Care Unit
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sixth Affiliated Hospital, Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, SanQing Jin, Professor, Sixth Affiliated Hospital, Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 2025ZSLYSC-630
Record Dates: First submitted 2025-11-18; First posted 2025-12-19 (Actual); Last update posted 2025-12-19 (Actual); Status verified 2025-12

CONDITIONS: Hypoxemia
Keywords: hypoxemia; oxygen concentration; atelectasis
MeSH Terms: conditions — Hypoxia; Pulmonary Atelectasis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group : 100% oxygen concentration (Active Comparator): Patients will inhale 100% oxygen from the end of surgery to tracheal extubation in the recovery period.
  Interventions: Other: 100% oxygen concentration inhaled
- Experimental group: 30% oxygen concentration (Experimental): Patients will inhale 30% oxygen from the end of surgery to extubation in the recovery period.
  Interventions: Other: 30% oxygen concentration inhaled

INTERVENTIONS:
Other: 100% oxygen concentration inhaled — Oxygen concentration inhaled from the end of surgery to tracheal extubation after general anesthesia in the recovery period is 100%.
  Arms: Control group : 100% oxygen concentration
Other: 30% oxygen concentration inhaled — Oxygen concentration inhaled from the end of surgery to tracheal extubation after general anesthesia in the recovery period is 30%.
  Arms: Experimental group: 30% oxygen concentration

SUMMARY:
Before extubation during the anesthesia recovery period, 100% oxygen is routinely inhaled to increase the oxygen reserves, maximizing the time window for anesthesiologists to adjust strategies when they encounter hypoxemia after extubation.

However, even inhaling a short period of pure oxygen can cause absorptive atelectasis, and may even impair the effectiveness of intraoperative protective ventilation measures continuing to post-operative period. The purpose of this study is to determine whether 30% oxygen before extubation after abdominal surgery could reduce hypoxemia incidence after extubation during the recovery period or not, compared to 100% oxygen. 590 patients scheduled to abdominal surgeries, will be randomly assigned to receive 30% or 100% oxygen concentration from the end of surgery to extubation after general anesthesia in the post-anesthesia care unit. The incidence of hypoxemia (SpO2 < 90%) from extubation to leaving the post-anesthesia care unit (PACU) is the primary outcome.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18-65 years old, scheduled for elective abdominal surgery in general anesthesia with endotracheal intubation; ASA I-III grade; cardiac function 1-2 grade; 18 kg/m2 < BMI < 28 kg/m2; Preoperative SpO2 ≥ 94% without oxygen supplementation at rest; pre-anesthesia assessment shows no difficult airway, no difficulty with mask ventilation, no difficulty in intubation during tracheal insertion, and no difficulty in extubation as expected.

Exclusion Criteria:

* Respiratory infection recently, or atelectasis, inflammation, fibrosis, or pleural effusion by chest CT preoperatively.

History thoracic surgery and fractures of the sternum or ribs, chest deformity, difficulty in raising both upper limbs, or scoliosis.

High risk of reflux aspiration. Severe hepatic or renal dysfunction (e.g., Child-Pugh class C liver disease, or requiring dialysis).

Limb movement disorders. Mask ventilation or intubation difficulty during anesthesia induction. Occurrence of severe allergy, massive bleeding, suspected pulmonary embolism, pulmonary edema, myocardial injury, or cardiopulmonary arrest during surgery.

Currently participating in other clinical studies, which may have an impact on this study.

Inability to cooperate well for mental disorder, or hypophrenia.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 590 (Estimated)
Dates: Start 2025-12-30 (Estimated); Primary Completion 2026-05-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Incidence of hypoxemia | At the day of surgery from tracheal extubation to leaving the post-anesthesia care unit

SECONDARY OUTCOMES:
Incidence of post operative pulmonary-related complications | Within 7 days after surgery
Incidence of severe hypoxemia | At the day of surgery from tracheal extubation to leaving the post-anesthesia care unit
Arterial partial pressure of oxygen (PaO2) | At the day of surgery after tracheal extubation in the post-anesthesia care unit
Score of lung ultrasound | At the day of surgery after tracheal extubation in the post-anesthesia care unit
  The score of lung ultrasound ranges from 0 to 36, and a higher score means a worse ventilation.
Area of atelectasis shown on chest CT | At the day of surgery after tracheal extubation
Number of patients unplanned transfers to the ICU | 30 days after surgery
Length of postoperative stay | At hospital discharge
Number of patients return to the hospital after discharge | 30 days after surgery
Number of deaths | 30 days after surgery
Number of patients with important organ disfunction after surgery, including arrhythmia, acute myocardial injury, heart failure, renal function injury, liver function injury, and cerebrovascular accident. | 30 days after surgery

CONTACTS AND LOCATIONS:
Locations (1):
- the Sixth Affiliated Hospital of Sun Yat-Sen University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No